CLINICAL TRIAL: NCT05141188
Title: Prevalence Of Extended Spectrum Beta Lactamase Producing Organisms In Urinary Tract Infections
Brief Title: Extended Spectrum Beta Lactamase Producing Organisms In Urinary Tract Infections
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mayada Shaaban Amin, Resident of Clinical and Chemical Pathology, Sohag University
Other Study IDs: Soh-Med-21-10-10
Record Dates: First submitted 2021-10-07; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urinary tract infection is among the most common nosocomial and community acquired infections. The Information on prevailing levels of antimicrobial resistance among common pathogens that associated with urinary tract infection is useful in making an appropriate choice of empiric therapy .Resistance to antibiotic treatment in patients with urinary tract infections (UTIs) is a representative example of the increasing problem of antimicrobial resistance. Extended-spectrum β-lactamases (ESBLs) has emerged as an important mechanism of resistance in Gram-negative bacteria.

DETAILED DESCRIPTION:
Urinary tract infection is among the most common nosocomial and community acquired infections. The Information on prevailing levels of antimicrobial resistance among common pathogens that associated with urinary tract infection is useful in making an appropriate choice of empiric therapy .

Resistance to antibiotic treatment in patients with urinary tract infections (UTIs) is a representative example of the increasing problem of antimicrobial resistance. Extended-spectrum β-lactamases (ESBLs) has emerged as an important mechanism of resistance in Gram-negative bacteria.

Bacterial production of extended-spectrum β-lactamases (ESBL) significantly reduces the efficacy of the most commonly used beta-lactam antibiotics for the empiric therapy of infections caused by putative Gram-negative .

Extended Spectrum Beta-Lactamase (ESBL) is derived from the mutated beta-lactamase enzyme, Beta-lactamase is an enzyme produced by bacteria that acts to inactivate beta-lactam class of antibiotics .

Extended Spectrum Beta-Lactamase is most commonly produced by the Enterobacteriaceae group, especially Escherichia coli and Klebsiella pneumonia.

ESBL-producing bacteria can also be resistant to the antibiotics class of aminoglycoside, fluoroquinolone, tetracycline, chloramphenicol, and sulfamethoxazole-trimethoprim.

The presence of ESBL-producing bacteria in an infection can result in treatment failure. Antibiotic resistance causes a decrease in the effectiveness of treatment, increases transmission of infection, increases mortality, and increases the cost of health care, while the discovery of new antibiotics is getting less and less

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted on a group of patients who are diagnosed that have urinary tract infections

Exclusion Criteria:

* The cases that do not give bacterial growth .

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted on all patients who are diagnosed that have urinary tract infections
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to indicate the spread of extended spectrum beta lactamase producing gram negative bacteria ( that isolated from the urine of patients with urinary tract infections based on their susceptibility to antimicrobial agents ) | through study completion, an average of 1 year
  This study will be conducted on a group of patients who are diagnosed that have urinary tract infections .
  * Methods of the study:
  Antibiotic susceptibility will be examined on disk diffusion test on Mueller-Hinton agar (MHA) . The zones of growth inhibition around each of the antibiotic disks are measured to the nearest millimeter
The aim of this study is to indicate the spread of extended spectrum beta lactamase producing gram negative bacteria ( that isolated from the urine of patients with urinary tract infections based on their susceptibility to antimicrobial agents ) | through study completion, an average of 1 year
  This study will be conducted on a group of patients who are diagnosed that have urinary tract infections .
  * Methods of the study:
  Antibiotic susceptibility will be performed by automated method Vitek -2 system that measured by minimal inhibitory concentration (MIC) .